CLINICAL TRIAL: NCT03099408
Title: A Pilot Study of Efficacy and Safety of Oral Metronidazole Versus Oral Metronidazole With Lactobacillus Vaginal Suppositories to Prevent the Recurrence of Bacterial Vaginosis
Brief Title: Oral Metronidazole With Lactobacillus Vaginal Suppositories to Prevent Recurrence of Bacterial Vaginosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Shangrong Fan, Profesor, Peking University Shenzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016PUSZH001
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Bacterial Vaginosis; Recurrence
Keywords: Recurrence; Lactobacillus Vaginal Suppositories
MeSH Terms: conditions — Vaginosis, Bacterial; Recurrence | interventions — Metronidazole; Lacteol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metronidazole Oral (Active Comparator): Metronidazole Oral
  Interventions: Drug: Metronidazole Oral
- "Metronidazole" and "Lactobacillus" (Active Comparator): "Metronidazole" and "Lactobacillus"
  Interventions: Drug: "Metronidazole" and "Lactobacillus"

INTERVENTIONS:
Drug: Metronidazole Oral — Oral metronidazole 400 mg BID for 7 days at first month.
  Arms: Metronidazole Oral
Drug: "Metronidazole" and "Lactobacillus" — Oral metronidazole metronidazole 400 mg BID for 7 days at first month and Lactobacillus vaginal suppositories for 10 days at first month,second month and third month.
  Arms: "Metronidazole" and "Lactobacillus"

SUMMARY:
We are trying to determine if Oral Metronidazole with Lactobacillus Vaginal Suppositories is better than Oral Metronidazole in Preventing the Recurrence of Bacterial Vaginosis

DETAILED DESCRIPTION:
Bacterial vaginosis (BV) is the most prevalent cause of symptomatic vaginal discharge in the U.S. and has been associated with complications including preterm delivery of infants, pelvic inflammatory disease (PID), urinary tract infections (UTI) and acquisition/transmission of sexually transmitted diseases (STDs) including human immunodeficiency virus (HIV).

Control of BV has been advocated as a means of decreasing the prevalence of these complications. However, the etiology of BV remains unknown and the current treatment regimens are inadequate in terms of initial cure and recurrence rates.

Based on currently national guidelines by using oral metronidazole 400 BID for 7 days, a high recurrence rate of BV were reported.

We hypothesize that the Oral Metronidazole with Lactobacillus Vaginal Suppositories is better than Oral Metronidazole in Preventing the Recurrence of Bacterial Vaginosis

ELIGIBILITY:
Inclusion Criteria:

* Women be at least 18 years of age
* Have symptoms of vaginal odor and or/discharge
* Meet the clinical (Amsel) criteria for BV
* Willing to participate in research

Exclusion Criteria:

* Presence of another vaginal infection or STD
* Allergy to metronidazole
* Pregnant or nursing
* Use of oral or intravaginal antibiotics within the past 2 weeks
* HIV or other chronic disease
* Inability to keep return appointments
* Contraindications for Lactobacillus Vaginal Suppositories（those without sexual history）

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Cure rate of BV | 4 weeks
  Nugent score

SECONDARY OUTCOMES:
Recurrence of BV | 12 weeks
  Nugent score
Recurrence of BV | 24 weeks
  Nugent score

CONTACTS AND LOCATIONS:
Overall Officials: Shangrong Fan, M.D., Principal Investigator — Peking University Shenzhen Hospital; Salvatore Giovanni Vitale, M.D., Principal Investigator — Department of Human Pathology in Adulthood and Childhood, University of Messina (Italy)
Locations (1):
- Dept Obstetrics and Gynecology, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No